CLINICAL TRIAL: NCT04044950
Title: A Phase II Study of Neoadjuvant E7 TCR T Cell Immunotherapy for Borderline Resectable and Unresectable Stage I HPV-Associated Oropharyngeal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was closed due to investigator discretion based on the lack of ability to recruit patients and research goals of the program.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 190130; 19-C-0130
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Papillomavirus Infections; Oropharyngeal Neoplasms
Keywords: Intratumoral Injection; Biomarkers; T Cell Receptor; Immunotherapy; Neoadjuvant therapy
MeSH Terms: conditions — Papillomavirus Infections; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Approximately 3x10^8 E7 TCR T cells (based on the number of disease sites the patient has) will be injected on day 0.
  Interventions: Biological: E7 TCR

INTERVENTIONS:
Biological: E7 TCR — The injection will be approximately 3x10^8 E7 TCR T cells, unless fewer cells are generated, at each site of organ involvement (i.e. primary tumor, palpable lymph node (s)) in approximately 1-2 mL of volume.

SUMMARY:
Background: Researchers have found a new way to treat cancer. The therapy used in this study is called E7 TCR T cell therapy. This therapy is a type of treatment in which a participant s T cells (a type of immune system white blood cell) are changed in the laboratory to attack cancer cells. This treatment might help people with human papilloma virus (HPV)-associated oropharyngeal cancer. Oropharyngeal cancer is a type of head and neck cancer that happens in the oropharynx (the part of the throat at the back of the mouth, including the soft palate, the base of the tongue and the tonsils). Certain types of the HPV virus can cause this kind of cancer and this study is looking at those cause by HPV-16.

Objective: The purpose of this study is to find out if injecting E7 TCR T cells directly into cancer tumor(s) can be done without delaying standard treatment for stage I oropharyngeal cancer, which may include surgery or radiation therapy with chemotherapy.

Eligibility: People aged 18 and older with borderline resectable or unresectable Stage I, HPV-16 associated oropharyngeal cancer.

Design: Participants will be screened with HLA typing (a blood test needed for eligibility) and HPV testing of the cancer tumor (to determine if the cancer is HPV-16 positive). A new biopsy may be needed if tumor from an outside location is not available for HPV testing. Eligible participants will come to the NIH campus to have a screening evaluation which will include physical exam, review of medical history and current medications, blood and heart tests, imaging (X-ray, CT scan, MRI or PET scan), and evaluation of participant s veins that are used for drawing blood.

If the participant is eligible for the study based on the screening evaluation, they will have a baseline evaluation prior to receiving the experimental treatment which may include additional laboratory or imaging tests. A biopsy of the primary tumor may be performed before getting the cell injection and approximately 4 weeks after the cell injection.

Participants will have a large IV catheter inserted into a vein to undergo a procedure called leukapheresis. Leukapheresis is the removal of the blood by a machine to collect specific white blood cells. The remaining blood is returned to the body. This procedure is needed to collect the cells that will be modified to target the cancer. The cells are grown in the lab and given back to the participant through an injection into the participant's tumor. It takes 11-15 days to grow the cells.

Once the cells are ready, participants will receive an injection of E7 TCR T cells directly into the primary tumor and any lymph nodes that can be seen or felt on physical exam. The injection will be done in the clinic or the operating room and may require general anesthesia. Participants will recover in the hospital until they are well enough to go home, which will be about 1-2 days after the cell injection.

Participants will have follow-up visits starting 2 weeks after cell injection. These will be visits to monitor the safety of the treatment and to evaluate the response of the cancer to the treatment. If the cancer appears to be growing at the 2-week visit, participants will go back to their local doctor for further care. If the cancer is not growing, participants will return for another follow-up visit 4 weeks after cell injection to see how the cancer is responding. Regardless of whether the cancer is shrinking or not, all participants will be referred to their home physician for further care after the 4-week visit.

After receiving cell therapy, participants will be followed on a long-term gene therapy protocol. Participants will have blood drawn periodically to test if the cells have grown or changed. These blood tests will take place immediately before the cells, and then at 3, 6, 12 months for the first year and then annually. These tests can be drawn locally and sent to the NIH. Participants will be asked to return to the NIH annually for a physical examination for 5 years after they receive the cell injection. If participants are not able, to return to the NIH annually, they may be contacted at home and asked to have records sent from their local doctor. After that time, participants will be asked to fill -out a questionnaire for the next ten years, for a total follow-up period of 15 years.

DETAILED DESCRIPTION:
Background:

* Human papillomavirus (HPV)+ oropharyngeal cancer is an increasingly common type of cancer that frequently affects young patients.
* Although the prognosis of early-stage cancer is favorable, the treatments can result in significant life-long morbidity.
* Neoadjuvant therapy is an active area of investigation. The goal of neoadjuvant therapy in this setting is to reduce the risk of disease recurrence and permit the study of de- intensified definitive treatment of early-stage disease.
* E7 TCR T cells have demonstrated safety and clinical activity in treatment-refractory metastatic HPV+ cancers.

Objectives:

- To determine the feasibility of intratumoral injection of E7 TCR T cells as neoadjuvant therapy for borderline resectable and unresectable stage I HPV+ oropharyngeal cancer.

Eligibility:

- Patients greater than or equal to 18 years of age with borderline resectable or unresectable stage I HPV+ oropharyngeal cancer.

Design:

* This is a phase II, single arm, feasibility study of neoadjuvant E7 TCR T cell therapy for borderline resectable and unresectable stage I HPV+ oropharyngeal cancer.
* Patients will receive intratumoral injection of E7 TCR T cells into the primary tumor and involved regional lymph nodes
* Patients will not receive a conditioning chemotherapy regimen or systemic aldesleukin
* Patients will be referred for definitive standard of care therapy following completion of protocol therapy

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed stage I (AJCC 8th edition) oropharyngeal squamous cell carcinoma that has not been treated.
* HPV16+ tumor and HLA-A*02:01+ HLA type (p16+ by THC and HLA-A*02 is also acceptable for enrollment but not for treatment).
* Borderline/marginally resectable or unresectable oropharyngeal cancer. Resectability will be determined by the referring physician and confirmed by otolaryngologists at the NTH (confirmation is not needed for enrollment but is required prior to treatment.
* Measurable disease by RECTST v1.1 criteria.
* Patient age greater than 18 years. Because no dosing or adverse event data are currently available on the use of E7 TCR T cells in patients <18 years of age, children are excluded from this study.
* ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
* Patients must have normal organ and marrow function as defined below:

  * leukocytes greater than or equal to 3,000/mcL
  * absolute neutrophil count greater than or equal to 1,500/mcL
  * platelets greater than or equal to 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance greater than or equal to 60 mL/min/1.73 m(2) for patients with creatinine levels above institutional normal (calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation).
* Women of child-bearing potential must have a negative pregnancy test. Women of child-bearing potential are defined as all women who are not post-menopausal or who have not had a hysterectomy. Postmenopausal will be defined as women over the age of 55 who have not had a menstrual period in at least 1 year.
* The effects of E7 TCR T cells on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (intrauterine device, hormonal or barrier method of birth control; abstinence, tubal ligation or vasectomy) prior to study entry and for up to 4 months after treatment. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Seronegative for HIV antibody. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment.
* Seronegative for hepatitis B antigen and hepatitis C antibody. If hepatitis C antibody test is positive, then the patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
* Must be willing to participate in Gene Therapy Long Term Follow-up Protocol (20-C-0051), which will follow patients for up to 15 years per Food and Drug Administration (FDA) requirements.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Patients who are receiving any other investigational agents.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations at the time of treatment that would limit compliance with study requirements.
* Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with E7 TCR T cells, breastfeeding should be discontinued if the mother is treated with E7 TCR T cells.
* Patients with any form of systemic immunodeficiency, including acquired deficiency such as HIV or primary immunodeficiency such as Severe Combined Immunodeficiency Disease, are ineligible. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the treatment.
* Patients on immunosuppressive drugs.
* Concurrent systemic steroid therapy if greater than the equivalent of 5 mg prednisone PO daily. Patients previously on steroids must be off steroids for four weeks prior to treatment.
* Patients with active cardiac ischemia or severe chronic obstructive pulmonary disease are not eligible.
* Patients with a second active invasive cancer are not eligible if it may confound assessment of response to the current therapy.
* Patients who do not have a physician to provide standard therapy post cellular treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
The fraction who achieve a success among those who receive E7 TCR T cell administration and who can be evaluated for the three feasibility criteria with 95% confidence intervals on the fraction reported as well. | 3 months
  The fraction who achieve a success will be determined and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Hinrichs, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-C-0130.html